CLINICAL TRIAL: NCT01114464
Title: Impact of Chemotherapy on Ovarian Reserve in Young Women With Breast Cancer
Acronym: Resova
Status: Terminated | Type: Observational
Why Stopped: end of normal study
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/09/06-J
Record Dates: First submitted 2010-04-28; First posted 2010-05-03 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Reserve
Keywords: Breast cancer; Ovarian reserve; Anti-Mullerian Hormone (AMH); Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- young women with breast cancer

SUMMARY:
The aim of this protocol is to study the deleterious impact of adjuvant chemotherapy or neoadjuvant chemotherapy on ovarian reserve in young women suffering from breast cancer. A new relevant ovarian reserve marker, serum Anti-Mullerian Hormone, will be used in order to evaluate precisely the impact of chemotherapy on ovaries during chemotherapy administrations and after during follow-up (24 months). This strategy offers 2 main advantages : no modification of the traditional care of patients (treatment, organisation, follow up …) and use of a non invasive marker (serum). The final objective is to give precise information to patients on their future fertility after remission.

ELIGIBILITY:
Inclusion Criteria:

* female 18-39 years
* suffering from breast cancer
* treated with adjuvant or neoadjuvant chemotherapy

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of adjuvant or neoadjuvant chemotherapy treatment on ovarian reserve for in situ breast cancer patients | 24 months
  Serum anti-Müllerian hormone concentration will be measured at each chemotherapy administration and 24 months follow-up after chemotherapy completion

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barrière, MD, Principal Investigator — Nantes University Hospital
Locations (11):
- France (11):
  - Institut Bergonié, Bordeaux
  - Centre François BACLESSE, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CRLC de Bourgogne Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre de Lutte Contre le Cancer Léon Bérard, Lyon
  - Centre Val d'Aurelle - Paul Lamarque, Montpellier
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre de Lutte Contre le Cancer Nantes Atlantique René Gauducheau, Saint-Herblain

REFERENCES:
- [Derived] Loubersac S, Chaillot M, Reignier A, Lefebvre T, Dezellus A, Colombel A, Barriere P, Masson D, Freour T. Serum androgen dynamics in young women aged 18-40 treated with chemotherapy for breast cancer: an observational, multicentric, prospective study in France. Hum Fertil (Camb). 2024 Dec;27(1):2350758. doi: 10.1080/14647273.2024.2350758. Epub 2024 Jul 3. PMID 38957151